CLINICAL TRIAL: NCT04410250
Title: Effect of Oral Hygienization in Newborn on Candida Spp Colonization and Child Behavior During Hygiene Habits
Brief Title: Effect of Oral Hygienization in Newborn on Candida Spp Colonization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3.568.480
Record Dates: First submitted 2019-09-23; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Newborns; Oral Hygiene; Candidiasis, Oral; Behavior
Keywords: Neonate.; Newborn.; Oral hygiene.; Oral health.; Candidiasis.
MeSH Terms: conditions — Candidiasis, Oral; Behavior; Candidiasis | interventions — Oral Hygiene

STUDY DESIGN:
Intervention Model Description: Sample Size in Brazil: 102
  Groups into which survey participants will be divided at this center:
  Group 1: 51 (Newborns whose parents will receive oral hygiene guidelines prior to tooth eruption) Group 2: 51 ( Newborns whose parents will be advised not to perform oral hygiene prior to tooth eruption.)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blindness The interventions will always be made by the same researcher and will not participate in the evaluations.
  Examiner 1 will be blinded to the group in which the examined children were allocated. Mothers will be advised not to disclose the group in which they were allocated during the evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral hygiene before tooth eruption (Active Comparator): The mothers of the newborns allocated to Group 1 will be instructed to clean the child's oral cavity by massaging the gingival rods with gauze and filtered water once a day at night.
  Following the eruption of the child's first tooth, mothers will be instructed to brush twice a day with fluoride toothpaste (1100 ppm fluoride) in a minimum amount, equivalent to one grain of raw rice, using the Fones technique. circular movements in the buccal and lingual faces of all teeth (FONES, 1934).
  Interventions: Behavioral: oral hygiene
- Absence of oral hygiene before tooth eruption (Experimental): The mothers of the newborns allocated to Group 2 will be advised not to perform any type of oral cavity cleaning of the newborn.
  Following the eruption of the child's first tooth, mothers will be instructed to brush twice a day with fluoride toothpaste (1100 ppm fluoride) in a minimum amount, equivalent to one grain of raw rice, using the Fones technique. circular movements in the buccal and lingual faces of all teeth (FONES, 1934).
  Interventions: Behavioral: oral hygiene

INTERVENTIONS:
Behavioral: oral hygiene — Mothers will be instructed on the oral hygiene of the newborn

SUMMARY:
Oral hygiene is one of the most accessible and well-known strategies for the prevention of dental caries. The benefits of this practice after tooth eruption are well established in the literature. Oral hygiene in newborns prior to tooth eruption is controversial, since there is a disagreement between the Dental and Pediatric Associations as to the optimal time to initiate oral hygiene in children and scientific studies in this regard have not yet been performed. Some of these associations recommend starting this practice from the eruption of the child's first tooth. Others recommend beginning the cleansing of the child's oral cavity from birth by cleaning the baby's gingival rollers and tongue. The aim of the present investigation will be to evaluate, through a randomized clinical trial, the influence of oral hygiene in newborns on Candida spp colonization. and on the child's behavior during oral hygiene after tooth eruption. Will be included in the study, pairs of mothers and babies born in the maternity of the Hospital Nossa Senhora da Saúde, in Diamantina, Minas Gerais, Brazil.

This will be a rehearsal Randomized clinical trial in which newborns will be allocated into 2 groups, namely:

* Newborns whose parents will receive guidelines for oral hygiene before tooth eruption (Group 1);
* Newborns whose parents will receive instructions not to perform oral hygiene before tooth eruption (Group 2).

The initial data collection will be performed one month after the child's birth and will include oral clinical examinations, saliva collection and questionnaires on the socio-environmental, economic and behavioral aspects of the child and his family. Initial oral clinical examinations will be performed to assess the presence of Candidiasis, and saliva collection will be performed to identify and quantification of Candida spp. These evaluations will be performed again every three months. From the eruption of the first deciduous tooth, the follow-up included an assessment of the baby's behavior during oral hygiene performed by the responsible. This evaluation will be made by the examiner using the Frankl scale and HBCD scale criteria. Statistical analysis will be performed using the Statistical Package for Social Science, version 23.0 and will include descriptive, bivariate and multivariate analyzes.

DETAILED DESCRIPTION:
Project presentation:

Primary Objective:

To evaluate the influence of oral hygiene of newborns before dental eruption on colonization by Candida spp. and about the baby's behavior during oral hygiene performed by parents after tooth eruption.

Secondary Objective:

To evaluate the influence of oral hygiene of newborns before tooth eruption on Candida spp colonization and occurrence of candidiasis during the follow-up period. To evaluate the influence of oral hygiene of newborns before tooth eruption on the its behavior during oral hygiene performed by parents after tooth eruption.

Proposed Methodology:

Study design: Randomized blinded clinical trial in edentulous newborns who will be screened in their first two days of life at the Maternity Hospital of Our Lady of Health in Diamantina, Minas Gerais. If mothers agree to participate with their child in the study, contact and address will be requested for further data collection that will be performed at the participants' homes.

Intervention Groups:

* 1. Mothers will be instructed to sanitize the newborn's oral cavity prior to tooth eruption by massaging the gingival rods with gauze and filtered water once a day at night. Following the eruption of the child's first tooth, mothers will be instructed to brush twice daily with fluoride toothpaste (1100 ppm fluoride) in a minimum amount, equivalent to one grain of raw rice, using the Fones technique .
* 2. Mothers will be advised not to perform any type of oral cavity cleaning of the newborn before tooth eruption. Following the eruption of the child's first tooth, mothers will be instructed to brush twice daily with fluoride toothpaste (1100 ppm fluoride) in a minimum amount, equivalent to one grain of raw rice, using the Fones technique .

The calculation of the sample size was obtained from Lee, Laboratory of Epidemiology and Statistics, using the calculation of estimation of two proportions and adopting the parameters proportion of cases (positive behavior during hygiene according to the Frankl Scale) among the exposed (children receiving oral hygiene before tooth eruption): 65% (unpublished data from a previous study by the research group); Confidence level (1 -) = 95%; (= 0.05 or 5%); Test power (1-) = 80%; Relative risk: 1.5; Newborns by group: 42; 9 newborns (20%) will be added to each group to compensate for possible losses. Thus, the sample required for the development of the study will be 51 newborns and their mothers in each of the groups.

The work team will be composed by the Researcher 1, Examiner 1 and Assistants. Prior to the start of the study, these researchers will undergo a training and calibration process according to the role of each team. A pilot study will be performed on 10% of the sample, and if no methodological changes are required, these children will be included in the main study. Randomization will be performed by allocating participants in both intervention groups through a computer-generated random number. Examiner 1 will be blind to the group in which the examined children were allocated and the mothers will be advised not to disclose the group in which they were allocated.

Data Collection and Follow-up Instruments:

Social, Environmental, Behavioral and Health Data Form general of children.

Registration form for colonization evaluation of Candida spp.

Through the identification and quantification of Candida spp. using CHROMagar Candida culture medium. This evaluation will be performed in the first month and at 4 months after the birth of the child. Form for registration of the child's oral clinical examination to record the presence and / or absence of Oral Candidiasis, and if present, its location. After the eruption of the first tooth the examiner will classify the child's behavior according to the Frankl Scale and HBCD Scale using the child's behavior record form that will be used for the period. follow-up at 1 month, 4 months, 7 months, 10 months and 13 months. The child's diet will be assessed through eating habits at all follow-up times through 24-hour dietary reminders using the multi-pass method.

Risks:

The risks inherent to the study are related to the awkwardness of the guardian during the clinical evaluations and / or examinations in the babies, as well as the possible discomfort of the child during the oral clinical examination. However, examiners will be prepared to identify any possible discomfort and minimize or disrupt the assessment if necessary. The application of questionnaires to those responsible will be performed in the presence of the same, in order to reduce their embarrassment. The information collected will be accessible only by members of research.

Benefits:

The benefits to patients will be oral health guidelines, follow-up of children by the examiner and, if necessary, referral for dental treatment. For health professionals, the research will provide scientific evidence and support for guidance to the population that will benefit from such recommendations with better care for children's oral health and consequent improved oral health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Newborns who do not yet have erupted teeth at the time of the first assessment (1 month after birth).
* Newborns whose mothers agree with their participation and that of their child in the study.

Exclusion Criteria:

* Newborns who present with systemic impairment at the time of the first evaluation (1 month after birth), such as physical, neurological, respiratory diseases, gastroesophageal reflux disease, among others that may alter the oral microbiota.

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-08-06 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Colonization of Candida spp. | First month after the birth of the child
  In the first month after the birth of the child, an initial oral clinical examination and saliva collection will be performed to evaluate Candida spp colonization. These two assessments will be performed at the child's own home.
Colonization of Candida spp. | Four months after the birth of the child
  Four months after the birth of the child, an initial oral clinical examination and saliva collection will be performed to evaluate Candida spp colonization. These two assessments will be performed at the child's own home.

SECONDARY OUTCOMES:
Baby Behavior During Oral Hygiene | Seven months after the birth of the child
  The examiner will rate their behavior according to the Frankl Scale. To assess the Frankl scale or the examiner used to classify the behavior of four behavioral categories: (1) definitely positive; (2) positive; (3) negative; (4) definitely negative.
Baby Behavior During Oral Hygiene | Seven months after the birth of the child
  The examiner will rate their behavior according to the HBCD Scale. For an assessment of behavior, an amendment to the HBCD Code , will also be used, with the following definitions: H - A child makes some movement of the head, hindering responsible execution, except movements muscle facial or jaw movements. B - A child moves some part of the body, tries to interrupt the procedure, except when requested by the guardian. C - The child cries, complains or recovering from the procedures. D - The child's behavior interrupts responsible action, causing a delay in the procedure for at least 5 continuous seconds. To be considered non-collaborative, the child must have at least one of the above changes.
Baby Behavior During Oral Hygiene | Ten months after the birth of the child
  The examiner will rate their behavior according to the Frankl Scale. To assess the Frankl scale or the examiner used to classify the behavior of four behavioral categories: (1) definitely positive; (2) positive; (3) negative; (4) definitely negative.
Baby Behavior During Oral Hygiene | Ten months after the birth of the child
  The examiner will rate their behavior according to the HBCD Scale. For an assessment of behavior, an amendment to the HBCD Code , will also be used, with the following definitions: H - A child makes some movement of the head, hindering responsible execution, except movements muscle facial or jaw movements. B - A child moves some part of the body, tries to interrupt the procedure, except when requested by the guardian. C - The child cries, complains or recovering from the procedures. D - The child's behavior interrupts responsible action, causing a delay in the procedure for at least 5 continuous seconds. To be considered non-collaborative, the child must have at least one of the above changes.
Baby Behavior During Oral Hygiene | Thirteen months after the birth of the child
  The examiner will rate their behavior according to the HBCD Scale. For an assessment of behavior, an amendment to the HBCD Code , will also be used, with the following definitions: H - A child makes some movement of the head, hindering responsible execution, except movements muscle facial or jaw movements. B - A child moves some part of the body, tries to interrupt the procedure, except when requested by the guardian. C - The child cries, complains or recovering from the procedures. D - The child's behavior interrupts responsible action, causing a delay in the procedure for at least 5 continuous seconds. To be considered non-collaborative, the child must have at least one of the above changes.
Baby Behavior During Oral Hygiene | Thirteen months after the birth of the child
  The examiner will rate their behavior according to the Frankl Scale. To assess the Frankl scale or the examiner used to classify the behavior of four behavioral categories: (1) definitely positive; (2) positive; (3) negative; (4) definitely negative.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Beatriz S Lopes, Graduated, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri
Locations (1):
- Ana Beatriz Silva Lopes, Diamantina, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No